CLINICAL TRIAL: NCT04181138
Title: Prospective Observational Study of Primary Sclerosing Cholangitis (PSC) in Children
Brief Title: Primary Sclerosing Cholangitis in Children
Status: Recruiting | Type: Observational
Sponsor: Arbor Research Collaborative for Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: PSC Study - ChiLDReN Network; 2U24DK062456 (NIH)
Record Dates: First submitted 2019-08-06; First posted 2019-11-29 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Primary Sclerosing Cholangitis; Liver Diseases; Cholangitis, Sclerosing
Keywords: Pediatric Liver Disease; Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, plasma, serum, PBMCs, stool, liver tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Primary sclerosing cholangitis (PSC) is a rare liver disease that damages the liver's bile ducts. Bile ducts are tiny tubes that carry bile from the liver to the small intestine. Bile is a liquid produced by the liver that helps us absorb and use the nutrients in the food we eat. In people with PSC, the bile backs up into the liver and will damage it, causing scarring of the liver.

The purposes of this study are to:

* Collect medical and other data to learn more about PSC, how it progresses, and identify factors that may cause the disease to progress more quickly.
* Ask questions about how PSC symptoms affect your child's life to learn more about its impact on your child's daily functioning
* Children with PSC who are seen at one of the participating clinical sites in the Childhood Liver Disease Research Network (ChiLDReN) will be asked to contribute information, DNA, and other specimens. The information and specimens will be available to investigators to carry out approved research aimed at learning more about the possible causes and long-term effects of PSC.

DETAILED DESCRIPTION:
Pediatric primary sclerosing cholangitis (PSC) is a rare autoimmune biliary fibrosing disease that leads to significant morbidity, the need for liver transplantation in ~50% of patients, and an increased risk for biliary and colorectal cancers in adulthood. The progression of the biliary disease in children is variable and risk factors associated with a more rapid progression of disease have not been adequately studied. Importantly, pediatric hepatologists have never previously collaborated with inflammatory bowel disease (IBD) specialists to rigorously explore interactions between colonic inflammation and liver disease. New non-invasive imaging modalities to measure fibrosis have not been explored in pediatric PSC. Furthermore, the impact that PSC has on the global functioning of children is not well understood, and likely underappreciated.

The natural history of pediatric PSC is poorly understood. This study aims to determine risk factors, including activity of co-existent IBD, associated with more rapid progression of disease, characterize the impact of PSC on global functioning, define the spectrum and prognostic value of biliary tract disease and liver fibrosis based on novel imaging techniques, and establish a biobank of specimens for future mechanistic studies aimed at discovering biomarkers pertaining to etiology and severity of PSC and novel mechanisms of immunopathogenesis of disease. This comprehensive observational and longitudinal study will delineate unique aspects of the natural history and severity of pediatric PSC and of associated IBD and provide necessary data for future therapeutic trials. It aims to provide a platform to discover and validate circulating and imaging biomarkers, which may serve as surrogate endpoints in future interventional studies.

ELIGIBILITY:
Inclusion Criteria:

Patients with the clinical diagnosis of large or small duct PSC made at any time prior to enrollment are screened for eligibility to participate in this prospective cohort study. The site PI will determine eligibility following review of MRCP or ERCP images with the site radiologist to confirm presence of an abnormal cholangiogram at the time of diagnosis of large duct PSC. Liver histopathology obtained at the time of diagnosis of small duct PSC will be reviewed with the site pathologist prior to enrollment.

Individuals must meet all of the Inclusion criteria in order to be eligible to participate in the study:

1. Aged 2 through 25 years at time of screening.
2. Diagnosis of large duct PSC based on review of cholangiogram by MRC, ERC, or intraoperative cholangiogram (IOC) by the site radiologist and interpreted to be consistent with PSC, based on one or more of the following:

   * Focal structuring of the bile duct(s)
   * Dominant stricture of the common bile duct
   * Saccular dilatation of bile duct(s)
   * Beaded appearance of bile duct(s)
   * Pruning appearance of the distal bile duct branches

   AND/OR
3. Diagnosis of small duct PSC based on review of liver histopathology by the site pathologist and interpreted to be compatible with PSC:

   * Probable small duct PSC: biopsy with ≥3 of 5 criteria: periductal edema, concentric inflammation, bile duct injury, ductular reaction, and neutrophils in bile ducts (cholangitis) OR...
   * Definitive small duct PSC: Periductal fibrosis/ "onion skinning" around interlobular bile ducts or smaller profiles
4. Stated willingness to comply with all study procedures and availability for the duration of the study.
5. Able to provide informed consent/assent

Participants for the imaging study are eligible if they are:

1. Aged 8 through 25 years at the time of screening
2. No absolute contraindication to MRI
3. No skin condition that could be aggravated by MREL
4. Meet all other eligibility criteria of the PSC Observational Study
5. For whom none of the exclusion criteria apply

Exclusion Criteria:

An individual who meets any of the following criteria at baseline will be excluded from participation in this study.

1. History of liver transplantation
2. History bone marrow transplantation
3. History of primary or acquired immunodeficiency predisposing to secondary sclerosing cholangitis, for instance: hyper-IgM syndrome, severe combined immunodeficiency (SCID) syndrome, common variable immunodeficiency (CVID) syndrome, cartilage hair hypoplasia syndrome, or HIV/AIDS
4. History of histiocytosis, including Langerhans cell histiocytosis (LCH), or hemophagocytic lymphohistiocytosis (HLH)
5. History of ischemic cholangitis
6. History of portal vein thrombosis with biliopathy, veno-occlusive disease, or abdominal radiation vasculopathy
7. History of recurrent pyogenic cholangitis
8. History of biliary tract surgery for cholecystolithiasis prior to cholangiogram/liver biopsy evaluated to determine enrollment
9. History of biliary tract surgery for choledochal cyst
10. History of hepatocellular carcinoma, or hepatoblastoma
11. History of surgical biliary trauma
12. History of congenital cytomegalovirus (CMV) hepatitis
13. History of Sickle Cell Disease
14. History of cystic fibrosis, biliary atresia, Caroli disease/congenital hepatic fibrosis, or progressive familial intrahepatic cholestasis type 3/MDR3 disease
15. History of cardiac hepatopathy.
16. History of metabolic disorders, including Wilson's disease, glycogen storage disorder, Alpha-1 Antitrypsin deficiency
17. Diagnosis of systemic lupus erythematosus (SLE)
18. Concurrent pregnancy at the time of enrollment -

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants are eligible for enrollment into the ChiLDReN PSC Study if they meet the inclusion criteria and if none of the exclusion criteria apply. Every effort will be made to enroll as diverse a patient population (racial, ethnic, sex, age, etc) as possible.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-12-30 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
To characterize the major phenotypes of PSC including patients with large duct or small duct disease, with and without Inflammatory Bowel Disease (IBD), and with and without Auto Immune Hepatitis (AIH) | up to 10 years
  Data will be collected on all phenotypes of PSC but attention is focused on how the intestinal inflammation and clinical activity of Inflammatory Bowel Disease (IBD) affect the progression of PSC, better classification of patients with features of Auto Immune Hepatitis (AIH), and the implications of bacterial cholangitis amongst all PSC phenotypes.
  Collection of retrospective clinical and laboratory data from the time of diagnosis of PSC and annual timepoints thereafter. Information regarding clinically important timepoints, laboratory data and FibroScan Liver Stiffness Measurements (LSM) are collected prospectively.
  Slides/images (if available) from each liver biopsy obtained at the time of diagnosis of PSC and thereafter and from the explanted liver recovered at the time of liver transplantation will undergo central review.
  Cholangiography results (MRCP, ERCP) will also undergo central review.

SECONDARY OUTCOMES:
To identify the symptoms of PSC in children and the affects of those symptoms on the functional health of children. | up to 10 years
  Identify deficits in the functional health of children with PSC and explore the association of these functional parameters with biochemical markers of liver disease severity and IBD activity. Symptoms and the impact the symptoms on the functional health of children is measured through the use of "Patient Reported Outcomes" and performance-based metrics.
  The burden of disease on the quality of life for children with PSC is measured utilizing the Peds-QL questionnaires (parent proxy and self-report). Child self-report: 8-12 years, and 13-18 years. Young adult self-report: 18-25 years. Parent proxy report: 2-4 years, 5-7 years, 8-12 years, and 13-17 years.
  Itch and fatigue identified as predominant symptoms in PSC are measured through the administration (at every visit) of the 5-D ITCH scale and the PedsQL multidimensional fatigue and PROMIS Sleep Scales.
  Frailty parameters in children with PSC are measured through the Fried frailty criteria at every visit.
Utilizing imaging modalities measuring liver fibrosis, and large duct injury to correlate with other markers of fibrosis and biliary injury and predict progression of disease. | up to 10 years
  The imaging modalities are utilized to explore the two pathophysiological processes of PSC, liver fibrosis and bile duct damage. Quantitative MRI techniques may be more sensitive to disease progression than standard clinical and laboratory tests, as the liver and bile ducts are being explored directly.
  All participants will undergo a liver stiffness measurement (LSM) at baseline and annually. In addition to the LSM, participants who are eligible (eligibility criteria are different than those for the overall study) will be asked to undergo a research MRI at the baseline, Year 1 and Year 5 visits.
Development of a repository for formalin fixed paraffin embedded (FFPE) liver biopsy tissue, serum, plasma, peripheral blood mononuclear cells (PBMCs), DNA and stool. | up to 10 years
  Samples of peripheral blood mononuclear cells (PBMC), serum, plasma, DNA and stool are collected from participants at baseline and serum/plasma will be collected annually. In addition, any liver tissue previously collected or collected for clinical purposes in the future will be analyzed along with the PBMC, serum, plasma, DNA and stool within future mechanistic ancillary studies related to the diagnostic/prognostic biomarkers, and genetic, immune and microbial theories of pathogenesis.

CONTACTS AND LOCATIONS:
Overall Officials: Cara Mack, MD, Study Chair — Medical College of Wisconsin-Milwaukee; Ed Doo, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); Katrina Loh, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); John Magee, MD, Principal Investigator — University of Michigan; Lisa Henn, PhD, Principal Investigator — Arbor Research Collaborative for Health
Locations (12):
- United States (11):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H Lurie Children's Hospital, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Cincinnati Children's Hospital Medical, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital (Baylor College of Medicine), Houston, Texas
  - The University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] Hirschfield GM, Karlsen TH, Lindor KD, Adams DH. Primary sclerosing cholangitis. Lancet. 2013 Nov 9;382(9904):1587-99. doi: 10.1016/S0140-6736(13)60096-3. Epub 2013 Jun 28. PMID 23810223
- [Background] Eaton JE, Talwalkar JA, Lazaridis KN, Gores GJ, Lindor KD. Pathogenesis of primary sclerosing cholangitis and advances in diagnosis and management. Gastroenterology. 2013 Sep;145(3):521-36. doi: 10.1053/j.gastro.2013.06.052. Epub 2013 Jul 1. PMID 23827861
- [Background] Bambha K, Kim WR, Talwalkar J, Torgerson H, Benson JT, Therneau TM, Loftus EV Jr, Yawn BP, Dickson ER, Melton LJ 3rd. Incidence, clinical spectrum, and outcomes of primary sclerosing cholangitis in a United States community. Gastroenterology. 2003 Nov;125(5):1364-9. doi: 10.1016/j.gastro.2003.07.011. PMID 14598252
- [Background] Deneau M, Jensen MK, Holmen J, Williams MS, Book LS, Guthery SL. Primary sclerosing cholangitis, autoimmune hepatitis, and overlap in Utah children: epidemiology and natural history. Hepatology. 2013 Oct;58(4):1392-400. doi: 10.1002/hep.26454. Epub 2013 Aug 13. PMID 23686586
- [Background] Toy E, Balasubramanian S, Selmi C, Li CS, Bowlus CL. The prevalence, incidence and natural history of primary sclerosing cholangitis in an ethnically diverse population. BMC Gastroenterol. 2011 Jul 18;11:83. doi: 10.1186/1471-230X-11-83. PMID 21767410
- [Background] Olsson R, Danielsson A, Jarnerot G, Lindstrom E, Loof L, Rolny P, Ryden BO, Tysk C, Wallerstedt S. Prevalence of primary sclerosing cholangitis in patients with ulcerative colitis. Gastroenterology. 1991 May;100(5 Pt 1):1319-23. PMID 2013375
- [Background] Ricciuto A, Kamath BM, Griffiths AM. The IBD and PSC Phenotypes of PSC-IBD. Curr Gastroenterol Rep. 2018 Mar 28;20(4):16. doi: 10.1007/s11894-018-0620-2. PMID 29594739
- [Background] Mieli-Vergani G, Vergani D, Baumann U, Czubkowski P, Debray D, Dezsofi A, Fischler B, Gupte G, Hierro L, Indolfi G, Jahnel J, Smets F, Verkade HJ, Hadzic N. Diagnosis and Management of Pediatric Autoimmune Liver Disease: ESPGHAN Hepatology Committee Position Statement. J Pediatr Gastroenterol Nutr. 2018 Feb;66(2):345-360. doi: 10.1097/MPG.0000000000001801. PMID 29356770
- [Background] Debray D, Pariente D, Urvoas E, Hadchouel M, Bernard O. Sclerosing cholangitis in children. J Pediatr. 1994 Jan;124(1):49-56. doi: 10.1016/s0022-3476(94)70253-5. PMID 8283375
- [Background] Smolka V, Karaskova E, Tkachyk O, Aiglova K, Ehrmann J, Michalkova K, Konecny M, Volejnikova J. Long-term follow-up of children and adolescents with primary sclerosing cholangitis and autoimmune sclerosing cholangitis. Hepatobiliary Pancreat Dis Int. 2016 Aug;15(4):412-8. doi: 10.1016/s1499-3872(16)60088-7. PMID 27498582
- [Background] Feldstein AE, Perrault J, El-Youssif M, Lindor KD, Freese DK, Angulo P. Primary sclerosing cholangitis in children: a long-term follow-up study. Hepatology. 2003 Jul;38(1):210-7. doi: 10.1053/jhep.2003.50289. PMID 12830004
- [Background] Miloh T, Arnon R, Shneider B, Suchy F, Kerkar N. A retrospective single-center review of primary sclerosing cholangitis in children. Clin Gastroenterol Hepatol. 2009 Feb;7(2):239-45. doi: 10.1016/j.cgh.2008.10.019. Epub 2008 Oct 30. PMID 19121649
- [Background] Valentino PL, Wiggins S, Harney S, Raza R, Lee CK, Jonas MM. The Natural History of Primary Sclerosing Cholangitis in Children: A Large Single-Center Longitudinal Cohort Study. J Pediatr Gastroenterol Nutr. 2016 Dec;63(6):603-609. doi: 10.1097/MPG.0000000000001368. PMID 27504812
- [Background] Wilschanski M, Chait P, Wade JA, Davis L, Corey M, St Louis P, Griffiths AM, Blendis LM, Moroz SP, Scully L, et al. Primary sclerosing cholangitis in 32 children: clinical, laboratory, and radiographic features, with survival analysis. Hepatology. 1995 Nov;22(5):1415-22. PMID 7590657
- See also: Childhood Liver Disease Research Network (ChiLDReN) website — https://childrennetwork.org/